CLINICAL TRIAL: NCT00312923
Title: Preliminary Study of Safety and Efficacy of Policosanol
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Barbara Swanson, Assistant Professor, Rush University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: R21AT003077-01 (NIH); R21AT003077-01 (NIH)
Record Dates: First submitted 2006-04-07; First posted 2006-04-11 (Estimated); Results first posted 2013-07-15 (Estimated); Last update posted 2013-07-26 (Estimated); Status verified 2013-07

CONDITIONS: Dyslipidemia; HIV Infections
Keywords: HIV; lipids; dyslipidemia; policosanol; treatment experienced
MeSH Terms: conditions — Dyslipidemias; HIV Infections | interventions — policosanol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Policosanol (Experimental): 20 mg daily of policosanol
  Interventions: Drug: Policosanol
- Placebo (Placebo Comparator): 20 mg of microcrystalline cellulose daily
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Drug: Policosanol — 20 mg of policosanol in capsular form daily
  Arms: Policosanol
Dietary Supplement: Placebo — Two capsules of 10 mg of microcrystalline cellulose daily
  Arms: Placebo

SUMMARY:
Lay Language Summary: High cholesterol levels are common in persons with HIV infection. However, conventional cholesterol-lowering medications may have harmful side effects when given to HIV-infected persons. Therefore, we plan to evaluate the safety and effectiveness of policosanol, a dietary supplement derived from sugar cane that has cholesterol-lowering properties, to lower cholesterol levels in persons with HIV infection. We hypothesize that policosanol will lower levels of LDL cholesterol ("bad" cholesterol) and raise levels of HDL cholesterol ("good" cholesterol).

DETAILED DESCRIPTION:
As per Brief Summary

ELIGIBILITY:
Inclusion Criteria:

CD4 count > 250 Plasma HIV RNA < 50,000 Currently receiving HAART age 18-60 total cholesterol between 200-240 or triglycerides between 150-400 or LDL cholesterol > 160

Exclusion Criteria:

kidney or liver disease current use of lipid-lowering drugs pregnancy lactation

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2005-09; Primary Completion 2009-07 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara A Swanson, DNSc, Principal Investigator — Rush University College of Nursing
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between April, 2006 and July, 2009 at three inner-city outpatient HIV/AIDS clinics located in a Chicago neighborhood that has been designated as medically underserved by the Health Resources Service Administration (HRSA).
Pre-assignment Details: A total of 176 participants were screened for eligibility and 54 were randomized and entered into the intent-to-treat analyses. Most of the ineligible participants did not meet the study's lipid criteria
Groups:
- Treatment Group: 20 mg daily of policosanol
  Policosanol : 20 mg of policosanol in capsular form daily
- Control Group: Placebo : Two capsules of 10 mg of microcrystalline cellulose daily
Period: Overall Study
Arm/Group | Treatment Group | Control Group
Started | 28 | 26
Completed | 19 | 20
Not Completed | 9 | 6

BASELINE CHARACTERISTICS:
Population: 54 eligible participants were randomized to the study arms. 39 participants completed the study. An intent-to-treat analysis was performed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Control Group | Total
Number analyzed (Participants) | 28 | 26 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 26 | 54
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 44.6 (.54) | 46.8 (6.56) | 44.67 (6.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 21 | 18 | 39
Region of Enrollment [Number; unit: participants]
  United States | 28 | 26 | 54

OUTCOME MEASURES:

1. Primary Outcome: LDL Cholesterol
Description: Low density lipoprotein cholesterol
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 27 | 27
mg/dl | 116.34 (37.75) | 118.84 (38.38)

2. Secondary Outcome: Triglycerides
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 27 | 27
mg/dl | 173.73 (200.39) | 186.69 (125.60)

ADVERSE EVENTS:
Arm/Group | Treatment Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
It is possible that other constituents underlie policosanol's lipid-lowering activity. One study found that triacontanol inhibited HMG-CoA reductase in rat liver cells. Triacontanol was not detected in either lot of policosanol used in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No